CLINICAL TRIAL: NCT02630407
Title: Early Post-op. Viscosupplementation After Primary Anterior Cruciate Ligament (ACL) Reconstruction: a Randomized, Placebo Controlled Trial
Brief Title: Early Viscosupplementation After ACL Reconstruction: a Randomized Controlled Trial
Acronym: HA-ACL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Federica Balboni, BScD, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rizzoli HA-ACL
Record Dates: First submitted 2015-11-30; First posted 2015-12-15 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Complete Tear, Knee, Anterior Cruciate Ligament
MeSH Terms: interventions — Viscosupplementation

STUDY DESIGN:
Intervention Model Description: injection of saline VS injection of Hyaluronic acid
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid group (Experimental): Single injection of 3 ml HA (product name: Hymovis, Fidia Spa, Padova, Italy) the day after ACL reconstruction (after drainage removal)
  Interventions: Biological: viscosupplementation
- Placebo group (Placebo Comparator): Single injection of 3 ml saline solution the day after ACL reconstruction (after drainage removal)
  Interventions: Other: Placebo group

INTERVENTIONS:
Biological: viscosupplementation — A single 3 ml hyaluronic acid (HA) injection (viscosupplementation) performed the day after ACL reconstruction, after drainage removal
  Arms: Hyaluronic acid group
Other: Placebo group — A single 3 ml saline injection performed the day after ACL reconstruction, after drainage removal
  Arms: Placebo group

SUMMARY:
The possibility of using an intra-articular agent such as hyaluronic acid (HA) to reduce the post-operative inflammatory stress on the knee joint, limiting the use of other pain-killers and promoting a faster recovery after ACL reconstruction, seems attractive.

The aim of the present double blind, placebo controlled study is to evaluate the effects, both in terms of pain control and functional recovery, provided by a single HA injection performed in the early postoperative phase after ACL reconstruction.

The day after the ACL reconstruction (which is performed with the same technique for all the patients enrolled), the patients were randomized to receive a single injection of HA or 3 ml of saline solution. The randomization list was kept in a dedicated office and the injecting physician contacted it to know the treatment allocation just before the injection, that was performed by a lateral parapatellar approach, after removing the drainages and after attempting aspiration to evacuate any eventual residual blood from the joint. In order to maintain the patient blind to the treatment, a surgical drape was placed to prevent him to see the injective procedure.

All patients will be evaluated at 15, 30, 60, 180 and 360 days after surgery by using the following tools: SF-36, IKDC subjective, VAS for pain, EQ-VAS for general Health Status and Tegner score. Also the trans-patellar circumference and active and passive ROM of both knees were registered at each follow-up evaluation.

DETAILED DESCRIPTION:
Viscosupplementation is an injective approach used in the orthopaedic practice to manage chondropathy and osteoarthritis (OA) in different joints. In the last decades, several products have been developed by biomedical industries, with different biochemical and physical properties, with the aim of providing the best and long-lasting beneficial effects in OA patients. The rational supporting the use of viscosupplementation is due both to its biomechanical and biological actions. First of all, hyaluronic acid (HA) exerts a lubricant effect improving the rheological properties of synovial fluid thus reducing the mechanical stresses within the joint that are responsible for the activation of nociceptors and further cartilage surface wear. Furthermore, HA binds to cellular receptors and further stimulates endogenous production of hyaluronan, other extracellular matrix components, and it also counteracts inflammatory molecules and proteases that are overexpressed in a diseased joint . In light of these features, HA could be considered an "intra-articular drug" which can act both as a pain killer and joint regulator agent. These properties could be theoretically exploited also for different clinical applications than a chronic disease like OA. In particular, viscosupplementation might play a beneficial role in restoring the overall joint homeostasis and might contribute to reduce pro-inflammatory stimuli after knee surgical procedures, thus reducing pain and accelerating functional recovery. Anterior cruciate ligament (ACL) reconstruction is one of the most common procedures in the field of sports medicine . It is common for patients to experience persistent knee swelling after the surgical procedure, and this increases pain and delays the start of the rehabilitation program, thus prolonging the times of full functional recovery. The possibility of using an intra-articular agent such as HA to reduce the post-operative inflammatory stress on the knee, limiting the use of other pain-killers and promoting a faster recovery after ACL reconstruction, seems therefore attractive.

The aim of the present double blind, placebo controlled randomized study is to evaluate the effects, both in terms of pain control and functional recovery, provided by a single HA injection performed in the early postoperative phase after ACL reconstruction.

The day after the ACL reconstruction (which is performed with the same technique for all the subjects enrolled), the patients were randomized to receive a single injection of HA or 3 ml of saline solution. The randomization list was kept in a dedicated office and the injecting physician contacted this office to know the treatment allocation just before the injection, that was performed by a lateral parapatellar approach, after removing the drainages and after attempting aspiration to evacuate any eventual residual blood from the joint. In order to maintain the patient blind to the treatment, a surgical drape was placed to prevent him to see the injective procedure.

All patients will be evaluated at 15, 30, 60, 180 and 360 days after surgery by using the following tools: SF-36, IKDC subjective, VAS for pain, EQ-VAS for general Health Status and Tegner score. Also the trans-patellar circumference and active and passive ROM of both knees were registered at each follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* chronic and symptomatic ACL tear requiring primary surgical reconstruction;
* age between 18 and 50 years;

Exclusion Criteria:

* concurrent articular lesion requiring surgical treatment (just isolated partial meniscectomy was permitted)
* axial mal-alignment in the index limb
* unhealthy contra-lateral knee (i.e. functional limitation or pain)
* concurrent rheumatic or metabolic disease
* alterations in the other joints of the index limb (e.g.: hip or ankle disease)
* previous ACL reconstruction in the index knee

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in IKDC (International Knee Documentation Committee) Subjective score | basal, 6 and 12 months post-op

SECONDARY OUTCOMES:
Change in Tegner Score | basal, 6 and 12 months
Transpatellar circumference trend | basal, 15, 30, 60, 180 days post op
Trend in Active and Passive Range of Motion (ROM) of the knee | basal, 15, 30, 60, 180 days post op
Change in VAS (Visual Analogue Scale) for general health status | basal, 15, 30, 60, 180 days post op
Change in VAS for pain | basal, 15, 30, 60, 180 days post op
Change in SF-36 (Short Form Health Survey) Score | basal, 6 and 12 months post-op
Adverse events report | 15 days
Adverse events report | 30 days
Adverse events report | 60 days
Adverse events report | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — II Clinic & Nano-biotechnology Lab, Rizzoli Orthopaedic Institute, Bologna, Italy
Locations (1):
- II Orthopaedic Clinic, Rizzoli Orthopaedic Institute, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Monticone M, Frizziero A, Rovere G, Vittadini F, Uliano D, LA Bruna S, Gatto R, Nava C, Leggero V, Masiero S. Hyaluronic acid intra-articular injection and exercise therapy: effects on pain and disability in subjects affected by lower limb joints osteoarthritis. A systematic review by the Italian Society of Physical and Rehabilitation Medicine (SIMFER). Eur J Phys Rehabil Med. 2016 Jun;52(3):389-99. Epub 2015 Sep 10. PMID 26365146
- [Background] Henrotin Y, Raman R, Richette P, Bard H, Jerosch J, Conrozier T, Chevalier X, Migliore A. Consensus statement on viscosupplementation with hyaluronic acid for the management of osteoarthritis. Semin Arthritis Rheum. 2015 Oct;45(2):140-9. doi: 10.1016/j.semarthrit.2015.04.011. Epub 2015 Apr 30. PMID 26094903
- [Background] Campbell KA, Erickson BJ, Saltzman BM, Mascarenhas R, Bach BR Jr, Cole BJ, Verma NN. Is Local Viscosupplementation Injection Clinically Superior to Other Therapies in the Treatment of Osteoarthritis of the Knee: A Systematic Review of Overlapping Meta-analyses. Arthroscopy. 2015 Oct;31(10):2036-45.e14. doi: 10.1016/j.arthro.2015.03.030. Epub 2015 May 19. PMID 25998016
- [Background] Filardo G, Di Matteo B, Di Martino A, Merli ML, Cenacchi A, Fornasari P, Marcacci M, Kon E. Platelet-Rich Plasma Intra-articular Knee Injections Show No Superiority Versus Viscosupplementation: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1575-82. doi: 10.1177/0363546515582027. Epub 2015 May 7. PMID 25952818
- [Background] Macdonald SA, Heard SM, Hiemstra LA, Buchko GM, Kerslake S, Sasyniuk TM. A comparison of pain scores and medication use in patients undergoing single-bundle or double-bundle anterior cruciate ligament reconstruction. Can J Surg. 2014 Jun;57(3):E98-104. doi: 10.1503/cjs.018612. PMID 24869623
- [Background] Braithwaite GJ, Daley MJ, Toledo-Velasquez D. Rheological and molecular weight comparisons of approved hyaluronic acid products - preliminary standards for establishing class III medical device equivalence. J Biomater Sci Polym Ed. 2016;27(3):235-46. doi: 10.1080/09205063.2015.1119035. Epub 2015 Dec 31. PMID 26569146
- [Background] Chau JY, Chan WL, Woo SB, Cheng SC, Wong TM, Wong TK, Yen CH, Wong K, Wong WC. Hyaluronic acid instillation following arthroscopic anterior cruciate ligament reconstruction: a double-blinded, randomised controlled study. J Orthop Surg (Hong Kong). 2012 Aug;20(2):162-5. doi: 10.1177/230949901202000205. PMID 22933671
- [Background] Huang MH, Yang RC, Chou PH. Preliminary effects of hyaluronic acid on early rehabilitation of patients with isolated anterior cruciate ligament reconstruction. Clin J Sport Med. 2007 Jul;17(4):242-50. doi: 10.1097/JSM.0b013e31812570fa. PMID 17620776
- [Derived] Di Martino A, Tentoni F, Di Matteo B, Cavicchioli A, Lo Presti M, Filardo G, Zaffagnini S, Marcacci M, Kon E. Early Viscosupplementation After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Am J Sports Med. 2016 Oct;44(10):2572-2578. doi: 10.1177/0363546516654909. Epub 2016 Jul 27. PMID 27466224